CLINICAL TRIAL: NCT07311863
Title: Study to Evaluate the Safety and Preliminary Efficacy of UGX202 Injection in Patients With Advanced Retinitis Pigmentosa
Brief Title: UGX202 Injection in Patients With Advanced Retinitis Pigmentosa
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Suzhou UgeneX Therapeutics Co., Ltd. (Other)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UGENEXIIT002
Record Dates: First submitted 2025-11-14; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Retinitis Pigmentosa (RP)
Keywords: UGX202; UGENEXIIT002; retinitis pigmentosa; RP; AAV
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose of UGX202 group (Experimental): UGX202, 4.2E+10 vg per eye, administered as a single intravitreal injection
  Interventions: Genetic: UGX202 injection
- High dose of UGX202 group (Experimental): UGX202, 1.2E+11 vg/eye, administered as a single intravitreal injection
  Interventions: Genetic: UGX202 injection

INTERVENTIONS:
Genetic: UGX202 injection — Comparison of different dosages of UGX202

SUMMARY:
The primary objective of this clinical trial is to evaluate the safety and tolerability of a single intravitreal injection of the gene therapy drug UGX202 in patients with advanced RP. The secondary objective is, to assess the preliminary efficacy of a single intravitreal injection of the gene therapy drug UGX202 in treating patients with advanced RP.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label investigator-initiated trial (IIT). It plans to enroll approximately 6 subjects with non-syndromic retinitis pigmentosa (RP) who have extremely low vision (the study eye is the eye with lower vision, and the best corrected visual acuity [BCVA] > logMAR 1.9).

The study drug is divided into two dose groups: low dose and high dose. A modified "3+3" dose escalation approach is adopted. The low-dose group (4.2E+10 vg/eye) is planned to include 3 subjects. First, 1 subject (sentinel) will be enrolled and observed for 28 days. If no dose-limiting toxicity (DLT) occurs, 2 more subjects (non-sentinel) will be enrolled and observed for 28 days. The second and third subjects will be enrolled with a 7-day interval.

The high-dose group (1.2E+11 vg/eye) is planned to include 3 subjects. Subjects in the high-dose group will be enrolled and administered the drug in sequence after passing the screening. There will be at least a 1-week interval between each subject. The timing of enrolling the full 3 subjects or stopping enrollment will be determined by the investigator's assessment of safety.All subjects will receive intravitreal injection of the study drug UGX202 after enrollment and will be followed up for 52 weeks to evaluate the safety, tolerability, and preliminary efficacy of UGX202.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent form (ICF).
* Age ≥18 years at ICF signing.
* Diagnosed as non-syndromic RP；
* BCVA > logMAR 1.9 (assessed by FrACT) in the study eye.
* Confirmation of preserved memory of visual experience
* Spherical equivalent between -9D and +6D.

Exclusion Criteria:

* Prior gene therapy in either eye.
* Received any interventional investigational drug within 90 days prior to screening.
* Any Study eye disease or systemic disease judged by the investigator to affect visual function assessment.
* Hypersensitivity to corticosteroids, intolerance to corticosteroid regimen, active concurrent infection contraindicating treatment.
* History or tendency of psychiatric disorders impacting safety and/or efficacy assessment.
* Any other factor deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | baseline to Day 3, Day 7, Week 2, Week 4, Week 6, Week 8, Week 12, Week 24, Week 36, Week 52
  From the time of administration of UGX202 injection until the 52nd week, based on the topical and systemic safety data, the incidence rates of AEs, TEAEs during treatment, TRAEs related to the study drug, TRAEs related to the study procedures, SAEs, TRSAEs related to the study drug, and TRSAEs related to the study procedures during the study period were summarized by the investigators, and the correlations between AEs and the study drug and study procedures were determined.
The average change in IOP | baseline to Day 3, Day 7, Week 2, Week 4, Week 6, Week 8, Week 12, Week 24, Week 36, Week 52
  The average change in IOP of the study eyes and non-study eyes from after treatment to the 52nd week compared to the baseline. The IOP was measured three times consecutively at each visit and the average value was taken.

SECONDARY OUTCOMES:
The changes in BCVA | baseline to Day 3, Day 7, Week 2, Week 4, Week 6, Week 8, Week 12, Week 24, Week 36, Week 52
  The changes in BCVA of the study eyes and non-study eyes at each follow-up visit compared to the baseline were evaluated. BCVA was assessed using the Freiburg Vision Test (FrACT) system. If the subjects had no light perception at the baseline: the proportion of subjects whose BCVA improved to having light perception after treatment was evaluated, and the change in their vision compared to the baseline was assessed;
The changes in the average stimulus threshold | baseline to Week 4, Week 12, Week 24, Week 52
  The changes in the average stimulus threshold measured by the full-field stimulus threshold test (FST) of the study eyes and/or non-study eyes at each follow-up visit compared to the baseline;
The changes in the visual function questionnaire (VFQ-25) scores | baseline to Day 3, Day 7, Week 2, Week 4, Week 6, Week 8, Week 12, Week 24, Week 36, Week 52
  The changes in the visual function questionnaire (VFQ-25) scores of the subjects at each follow-up visit after the treatment compared to the baseline.

OTHER OUTCOMES:
The change in Latency of N2, latency of P2, N2-P2 amplitude difference will be evaluated in VEP | Baseline, week4, week 8, week 12, week 24, week 52/EoS
  Latency of N2, latency of P2, N2-P2 amplitude difference will be evaluated in VEP both in the study eye and non-study eyes at each visits compared with baseline.
The change in dark-adapted 0.01 ERG, dark- adapted 3.0 ERG, dark-adapted 30.0 ERG and light-adapted 3.0 ERG | Baseline, week4, week 8, week 12, week 24, week 52/EoS
  Dark-adapted 0.01 ERG, dark- adapted 3.0 ERG, dark-adapted 30.0 ERG and light-adapted 3.0 ERG will be evaluated in electroretinogram both in the study eye and non-study eyes at each visits compared with baseline.
Change of mean defect (MD) in the visual fields | Baseline, week 24, week 52/EoS
  Change of mean defect (MD) in the visual fields of the study eyes and non-study eyes
Change of visual field index (VFI) in the visual fields | Baseline, week 24, week 52/EoS
  Change of visual field index (VFI) in the visual fields of the study eyes and non-study eyes
The benefit outcomes of patients with retinitis pigmentosa (RP) of different genotypes in either best-corrected visual acuity (BCVA) or the multi-luminance mobility test (MLMT) | Baseline
  The benefit outcomes of patients with retinitis pigmentosa (RP) of different genotypes either in best-corrected visual acuity (BCVA) or the multi-luminance mobilitytest (MLMT), and will conduct correlation the above analysis between factors.
Changes in the scores of MLMT | Baseline，week4， week 8, week 12, week 24, week 52/EoS
  Changes in the scores of multi-luminance mobility test (MLMT)
Change of Color Vision Test score | Baseline, week4, week 12, week 24, week 52/EoS
  Color vision test will be conducted to patients' assess judgment and discrimination abilities for different channels, with comparisons of the changes in scores at different study visits related to the baseline scores.
Titer of viral vector DNA detected in blood, tears, and urine | Baseline，Day3， Day7, week2, week 12, week 24, week 52/EoS
  Detection of viral vector DNA in blood, tears, and urine
Number of participants with positive Anti-drug antibodies(ADA) and neutralizing antibodies(Nab) | Baseline, week2, week4, week 12, week 24, week 36, week 52/EoS
  From the time of administration of UGX202 injection until the 52nd cycle, the detection of anti-drug antibodies (ADA) and neutralizing antibodies (Nab) for the viral vector capsid protein was carried out.
Number of participants with positive anti-target photosensitive protein | Baseline, week2, week4, week 12, week 24, week 36, week 52/EoS
  From the time of administration of UGX202 injection until the 52nd cycle, ADA (anti-target photosensitive protein) detection was conducted.
Concentration of T-cell immune responses against the viral vector capsid protein and the target photosensitive protein. | Baseline, week 12, week 24
  From the time of UGX202 injection treatment until the 52nd cycle, ELISpot was used to detect T-cell immune responses against the viral vector capsid protein and the target photosensitive protein.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No